CLINICAL TRIAL: NCT00776620
Title: A Relative Bioavailability Study of Glimepiride 1 MG Tablets Under Fed Conditions
Brief Title: Bioequivalence Study of Glimepiride 1mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr Tausif Monif, Ranbaxy Research laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10381502
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Glimepiride Tablets
MeSH Terms: interventions — glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Glimepiride 1 MG Tablets of Ranbaxy
  Interventions: Drug: Glimepiride 1mg Tablets
- 2 (Active Comparator): AMARYL® 1 mg tablets
  Interventions: Drug: Glimepiride 1mg Tablets

INTERVENTIONS:
Drug: Glimepiride 1mg Tablets

SUMMARY:
The objective of this study is to compare the relative bioavailability of glimepiride 1 mg tablets (manufactured by Ranbaxy Laboratories Limited) with that of AMARYL® 1 mg tablets (following a single oral dose (1 x 1 mg tablet) in healthy, adult subjects under fed conditions.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioequivalence study on glimepiride comparing glimepiride 1mg tablets of Ranbaxy laboratories limited with Amaryl 1mg tablets of in healthy, adult, human, subjects under fed conditions.

Thirty-two (32) subjects were recruited for this study and all subjects were healthy adults. Thirty-two (32) subjects began the study, and thirty-two (32) completed the clinical portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Source of Subjects: Non-institutionalized subjects consisting of members of the community at large.
* Characterization of Study Group.

  * All subjects selected for this study will be at least 18 years of age.
  * Each subject shall be given a general physical examination within 28 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.
* Each female subject will be given a serum pregnancy test as part of the pre-study screening process. At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements. Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.
* Clinical laboratory measurements will include the following:

  * Hematology: hemoglobin, hematocrit, red blood cell count, platelets, and white blood cell count (with differential).
  * Clinical Chemistry: creatinine, BUN, glucose, SGOT/AST, SGPT/ALT, bilirubin, and alkaline phosphatase.
  * Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells.
  * HIV Screen:(pre-study only)
  * Hepatitis-B, C Screen:(pre-study only)
  * Drugs of Abuse Screen:pre-study and at check-in each study period
* Subjects will be selected if all above are normal.
* Electrocardiograms of all participating subjects will be recorded before initiation of the study and filed with each subject's case report forms.

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption I,(during past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease,tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study. d. All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate.
* Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g.condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate.
* Subjects who have used implanted or injected hormonal contraceptives anytime during the 6 months prior to study dosing, or used oral hormonal contraceptives within 14 days before dosing will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or Inconclusive results will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-07; Primary Completion 2003-08 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html